CLINICAL TRIAL: NCT02621866
Title: A Trial of Daily Ultraviolet Therapy to Reduce Cardiovascular Risk Factors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PG/15/23/31362
Record Dates: First submitted 2015-06-25; First posted 2015-12-04 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2019-09

CONDITIONS: Hypertension
Keywords: hypertension; ultraviolet
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): UVA irradiation.
  Interventions: Device: Ultraviolet A radiation
- Sham UVA irradiation (Sham Comparator)
  Interventions: Device: Sham irradiation

INTERVENTIONS:
Device: Ultraviolet A radiation — Twice daily with 10 Joules/cm2. Half body (one side) with Waldmann 100L phototherapy lamp fitted with UVA bulbs (main emission 320-410nm)
  Other Names: UVA
  Arms: Active
Device: Sham irradiation — As active, but lamps to be shielded with Amber 81 museum film which prevents transmission of <500nm, but permits visible light to pass.
  Other Names: Screened UVA lamp
  Arms: Sham UVA irradiation

SUMMARY:
The investigators have shown that a single dose of ultraviolet irradiation (as found in sunlight) will lower blood pressure for around one hour. They are now testing whether daily UVA for two weeks will produce a sustained fall in BP in patients with high blood pressure.

They will also measure the effect of daily UVA on other cardiovascular risk factors.

DETAILED DESCRIPTION:
Epidemiological studies suggest that sunlight reduces all cause mortality, and particularly cardiovascular mortality.

The investigators have previously shown vasodilatation and a transient fall in blood pressure following irradiation of human volunteers with 2 standard erythemal doses of UVA radiation. This was independent of vitamin D and temperature rise and correlated with a nitric oxide synthase independent mobilisation of NO stores from the skin to the systemic circulation.

In this randomised, sham-controlled, cross-over double blind study, they will measure whether twice daily UVA administration can produce a sustained fall in BP and other cardiovascular risk factors in a cohort of pre-hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Pre-hypertensives (BP 120-139/80-89).
* Fitzpatrick skin types 2 and above (i.e. the ability to tan)

Exclusion Criteria:

* History of skin cancer.
* Fitzpatrick type 1 skin (always burns, never tans).
* Red hair.
* Family history of melanoma in first degree relative.
* Atypical naevus syndrome.
* Planned holiday or foreign travel during and for 4 weeks before the period of the study.
* Concurrent administration of:

  * anti-hypertensive medication,
  * photosensitising medication,
  * systemic immunosuppressive medication.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
24 hour ambulatory blood pressure measurement | Two weeks
  Before and after active and sham intervention period. Subjects will wear a 24 hour ambulatory blood pressure monitor for the 24 hour period before and after each 2 week intervention period. Change in 24 hour ambulatory blood pressure measurement will be the outcome measure.

SECONDARY OUTCOMES:
Blood pressure | Two weeks
  Measured with a mercury sphygmomanometer in clinical research facility. Change in blood pressure between the before and after measurements in the active and sham intervention.
Heart rate | Two weeks
  Change in heart rate between the before and after measurements of the active and sham intervention. This will be measured manually in clinical research facility before and after active or sham intervention period.
Body Mass Index | Two weeks
  Change in body mass index measured in clinical research facility before and after active and sham intervention period
Waist-Hip Ratio | Two weeks
  Change in waist-hip ratio. Measured in clinical research facility before and after active or sham intervention period
Lipid profile | Two weeks
  Change in lipid profile. Blood will be taken in the clinical research facility before and after active and sham intervention period. Analysis will be performed by the core specialist assay service at the adjacent Queens Medical Research Institute of the University of Edinburgh. Lipids are measured as a continuous variable.
Adipokine profile | Two weeks
  Change in adipokine profile. Blood will be taken in the clinical research facility before and after active and sham intervention period. Analysis will be performed by the core specialist assay service at the adjacent Queens Medical Research Institute of the University of Edinburgh. Adipokines are measured as a continuous variable.
Glucose tolerance test | Two weeks
  The standard National Health Service Lothian Glucose Tolerance Test protocol will be carried out and changes in outcome measures recorded. These will be the fasting glucose and the two hour glucose level. Both are continuous variables.
  Phlebotomy and glucose administration wil be performed in the clinical research facility before and after active and sham intervention period
HbA1c (glycosylated haemoglobin) | Two weeks
  Change in glycosylated haemoglobin level. Blood will be taken in the clinical research facility before and after active and sham intervention period. Analysis will be performed by the core specialist assay service at the adjacent Queens Medical Research Institute of the University of Edinburgh. Glycosylated haemoglobin is measured as a continuous variable.
Fasting insulin level | Two weeks
  Change in fasting insulin level. Fasting blood will be taken in the clinical research facility before and after active and sham intervention period. Analysis will be performed by the core specialist assay service at the adjacent Queens Medical Research Institute of the University of Edinburgh. Insulin levels are measured as a continuous variable.
Bio-impedance for body fat | Two weeks
  Changes in body fat levels. These are measured in clinical research facility before and after active or sham intervention period. This is a continuous variable.
Serum Vitamin D level | Two weeks
  Changes in serum Vitamin D level. This is a continuous variable. Blood will be taken in the clinical research facility before and after active or sham intervention period. Analysis will be performed by the core specialist assay service at the adjacent Queens Medical Research Institute of the University of Edinburgh.
Adaptive pigmentation | Two weeks
  Changes in pigmentation. Measured in clinical research facility before and after active or sham intervention period. Colour will be measured on UV exposed back skin using a chromameter and the L*a*b*score. This is a continuous variable.
Mood | Two weeks
  Changes in mood. Patients will complete a mood questionnaire in the clinical research facility at the appointment before and after the active or sham intervention period. This is a continuous variable.
Physical activity level- composite measure. | Two weeks
  Differences in activity levels will be compared between active, sham and washout periods. A composite measure derived from the peak, mean, and overall activity will be recorded. Overall activity will be calculated as area under the curve over the measurement period. Activity will be measured as movement, recorded by continually worn actiwatches (movement monitors) throughout the duration of the study. These will be set to record movement in 1 minute epochs.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Weller, MD FRCP, Principal Investigator — University of Edinburgh
Locations (1):
- Clinical Research Centre and Pharmacology Unit, Western General Hospital, Edinburgh, United Kingdom

REFERENCES:
- [Result] Liu D, Fernandez BO, Hamilton A, Lang NN, Gallagher JMC, Newby DE, Feelisch M, Weller RB. UVA irradiation of human skin vasodilates arterial vasculature and lowers blood pressure independently of nitric oxide synthase. J Invest Dermatol. 2014 Jul;134(7):1839-1846. doi: 10.1038/jid.2014.27. Epub 2014 Jan 20. PMID 24445737